CLINICAL TRIAL: NCT03682640
Title: Azithromycin Insulin Diet Intervention Trial in Type 1 Diabetes
Acronym: AIDIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIDIT
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus; Metabolic Disease; Glucose Metabolism Disorders; Endocrine System Diseases; Juvenile Diabetes; Insulin Dependent Diabetes; Type 1 Diabetes Mellitus; Inflammation; Diet Modification
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Metabolic Diseases; Glucose Metabolism Disorders; Endocrine System Diseases; Inflammation | interventions — Azithromycin; Insulin Lispro

STUDY DESIGN:
Intervention Model Description: The study is a 2-arm, randomized, open, clinical trial comparing the AIDIT protocol with treatment as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AIDIT protocol (Experimental): Treatment as usual with the addition of:
  i) Azithromycin Monohydrate, three times a week (≥ 48 h between doses) during 52 weeks. 500 mg if body weight ≥ 30 kg, 250 mg if body weight < 30 kg.
  ii) Extra intensive insulin treatment periods for maximum beta-cell rest with Insulin lispro (Sanofi). This treatment will be given i.v. for one episode of 72 hours in the first week after inclusion and s.c. on seven 6-8 h occasions during the study year. The dose will be individually titrated to reach target blood glucose 4.0±0.5 mmol/L.
  ii) Dietician support; Extra advice and support from the study dietician within the first week after randomization and after 1.5 and 4 months.
  Interventions: Drug: Azithromycin Monohydrate; Drug: Insulin Lispro; Behavioral: Dietician support
- Control (No Intervention): Patients will receive treatment as usual (TAU). All patients will receive standard therapeutic treatment consisting of insulin replacement with insulin analogues aiming for normoglycemia from diagnosis. Rapid acting insulin analogue will be administered via insulin pump (continuous subcutaneous infusion) with access to insulin injections in case of malfunction in the pump system.

INTERVENTIONS:
Drug: Azithromycin Monohydrate — Azithromycin Monohydrate tablet (Azithromycin Sandoz) or oral suspension (Azithromax).
  Other Names: Azithromycin Sandoz; Azithromax
  Arms: AIDIT protocol
Drug: Insulin Lispro — Solution for intravenous or subcutaneous use
  Other Names: Insulin lispro Sanofi
  Arms: AIDIT protocol
Behavioral: Dietician support — Dietary advice
  Arms: AIDIT protocol

SUMMARY:
Increasing evidences suggest that infections are important etiological factors for the development of Type 1 Diabetes (T1D). The overall hypothesis of the study is that the treatment of children, during the first year after diagnosis of T1D with Azithromycin, combined with repeated episodes of intensified insulin treatment to induce maximal beta-cell rest, and dietician support to promote dietary habits that minimize the likelihood of bacterial reflux from the duodenum to the pancreatic duct, will lead to preservation of beta cell function.

This trial will examine whether the AIDIT protocol initiated within one week from diagnosis could preserve insulin production in children with Type 1 Diabetes.

DETAILED DESCRIPTION:
The study is a 2-arm, randomized, open, single center, clinical trial. Eligible patients with type 1 diabetes will be randomized to the AIDIT protocol or treatment as usual (TAU).

All patients diagnosed with T1D and included in the study will receive standard of care. In addition, the AIDIT protocol will include 1) treatment with Azithromycin for 52 weeks using a protocol for children with cystic fibrosis, 2) repeated treatments with intensified supervised high dose insulin infusion, and 3) extra advice and support from the study dietician.

1. Azithromycin Azithromycin will be administered orally. Azithromycin will be given three times per week for 52 weeks. The dose will be 500 mg for children with body weight ≥ 30 kg and 250 mg if body weight < 30 kg.
2. Intensified supervised high dose insulin infusions Participants will, in addition to Azithromycin, also be subjected to intensified anti-diabetic treatment to achieve increased beta-cell rest. This will be achieved by insulin lispro given as a supervised iv infusion for 72 hours within one week of diagnosis and by subcutaneous infusion 6-8 hours during one day in study week 5, 9, 13, 17 (±1 week) and 25, 34, 43 (±2 weeks) after inclusion. The intensified treatments will aim to target a blood glucose level of 4.0 ± 0.5 mmol/l. The efficacy of the intended maximal beta cell rest will be evaluated by measurement of plasma glucose and endogenous C-peptide. If C-peptide remains positive during the supervised infusion of insulin lispro this will be interpreted as that the insulin dose needs to be increased at the next treatment occasion to achieve beta-cell rest.
3. Dietician support Participants will receive extra advice and support from the study dietician within the first week after randomization, and after 7 and 17 weeks. Personalized nutritional advice on intake of carbohydrates, fat and protein based on four-day food records will be given to in order to reduce insulin resistance and insulin need in accordance with ISPAD guidelines. By giving nutritional advices on less volume of the meals, especially of the fluid (maximum 300 ml per meal), and by trying to extend the meal time to at least 20 minutes, the reflux into ductus pancreaticus might be reduced.

All patients will be offered an examination of their pancreas with MRI at 0 and 12 months after inclusion. In addition, plasma samples taken at inclusion and after 1.5 and 12 months will be analysed for the presence of cell-free DNA indicating ongoing cell destruction. Cell-specific methylation patterns of this cell-free DNA will be analysed to determine cell-type specific cell death.

The effect of the addition of treatment according to the AIDIT protocol will be evaluated with a Mixed Meal Tolerance Test (MMTT) to explore the effect on preservation of beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed Type 1 Diabetes. First injection of insulin maximum ten days prior to inclusion.
2. Must be willing and capable of taking the study drugs, perform tests and follow up as described as judged by the investigator.
3. Signed informed consent and expected cooperation of the patients for the treatment and follow up.
4. Aged 6.00 -15.99 years at inclusion.
5. Females of childbearing potential must agree to avoid pregnancy during the study period (by abstinence from heterosexual intercourse, or by hormonal or barrier contraception) and have a negative urine pregnancy test.

Exclusion Criteria:

1. Other diabetes diagnosis than Type 1 diabetes as judged by the investigator
2. Severe ketoacidosis (DKA) with lowest pH <7.1 within 36 hours from diagnosis.
3. Treatment with any oral or injected anti-diabetic medications other than insulin
4. Significantly abnormal haematology results at screening.
5. Participation in other clinical trials with a new chemical entity within the previous 3 months.
6. Obesity at diagnosis (Iso-BMI ≥ 30 kg/m2 according to http://www.rikshandboken-bhv.se).
7. Other autoimmune disease present at inclusion that in the opinion of the investigator would interfere with the study protocol.
8. Celiac disease present at diagnosis.
9. Treatment with medication known to affect glucohomeostasis, i.e. glucocorticoids (inhaled, nasal or skin topic will be accepted), statins, ACE inhibitors.
10. Pregnancy or lactation
11. Known gastro-intestinal malabsorption disorders
12. Abnormalities in ECG or known cardiac disease
13. Known hearing defects
14. Known hypersensitivity to penicillin
15. Inability or unwillingness to comply with the provisions of this protocol
16. Presence of serious disease or condition in patient or family, which in the opinion of the investigator makes the patient non-eligible for the study.
17. Known renal or hepatic impairment

Ages: 72 Months to 192 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Stimulated C-peptide during an MMTT | 12 months after inclusion
  Residual insulin secretion measured by mixed meal tolerance test (MMTT) stimulated C-peptide two-hour under the curve profile measured one year after study inclusion.

SECONDARY OUTCOMES:
>60% of time in target blood glucose levels | two weeks in the 12th month after initiation of the study treatment
  Proportion of subjects with time in target 3.9-7.8 mmol/L ≥ 60% and with a glycaemic variability expressed as standard deviation < 2 mmol/L according to continuous glucose monitoring during two weeks in the 12th month after initiation of the study treatment.
Time in target blood glucose levels | 30 days in the 12th month after initiation of the study treatment
  Time in target (3.9-7.8 mmol/L) during 30 days in the 12th month after initiation of the study treatment.
Time in range blood glucose levels | 30 days in the 12th month after initiation of the study treatment
  Time in range (3.9-10 mmol/L) during 30 days in the 12th month after initiation of the study treatment.
Insulin dose | 30 days in the 12th month after initiation of the study treatment
  Mean daily insulin dosage per kilo bodyweight during 30 days in the 12th month after initiation of the study treatment.
HbA1c levels | 12 months
  HbA1c at 12 months after study initiation
Hypoglycaemic events | From study start to 12 months
  Number of severe hypoglycaemic events (hypoglycaemia level 3) during the study year.
Time in hypoglycemic range | 30 days in the 12th month
  Time in hypoglycaemic range level 1 and 2 (<3.9 mmol/l and <3.0 mmol/l) respectively in CGM registrations during 30 days in the 12th month after initiation of the study treatment.
IDAA1c | 12 months
  Insulin-dose-adjusted HbA1c (IDAA1c) 12 months after study initiation
Pro-insulin/c-peptide | 12 months
  Pro-insulin/c-peptide ratio in serum 12 months after study initiation
Pancreas inflammation | 12 months
  Inflammation in the pancreas measured by contrast enhanced MRI at 12 months after initiation of the study
QoL | 12 months
  Health related Quality of Life; Varni PedsQL, Generic and Diabetes specific questionnaire, by child and proxy (parents or other caregivers) at study start and 12 months after study initiation.
Gastrointestinal symptoms | 12 months
  Questionnaire on gastrointestinal symptoms: "The gastrointestinal symptom rating scale" (GSRS) at study start and 12 months after study initiation .
Time spent eating | 12 months
  Average time spent eating at meals during four days in the 12th month after initiation of the study treatment.
Intake of saturated fat | four days in the 12th month
  Intake of saturated fat (E% and if the child reaches Nordic Nutritional Recommendations, NNR) during four days in the 12th month after initiation of the study treatment.
Intake of fruit | four days in the 12th month
  Intake of fruit and vegetables (g/day and if the child reaches NNR) during four days in the 12th month after initiation of the study treatment.
Intake of macronutrients | four days in the 12th month
  Intake of macronutrients (E% and g/day) during four days in the 12th month after initiation of the study treatment.
Intake of fibre | four days in the 12th month
  Intake of fibre (g/day and if the child reaches NNR) during four days in the 12th month after initiation of the study treatment.
Physical activity measured with accelerometer | 6 months
  Physical activity registered with accelerometer during one week in the 6th month after initiation of the study treatment.
Physical activity measured with accelerometer | 12 months
  Physical activity registered with accelerometer during one week in the 12th month after initiation of the study treatment.
Oral microbiome | 12 months
  The oral microbiome at 12 months after study initiation.
Change in stimulated C-peptide | change from 6 weeks to 12 months after initiation of study treatment
  Change in stimulated c-peptide two-hour under the curve profile from 6 weeks to 12 months after initiation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gun Forsander, MD, PhD, Principal Investigator — The Queen Silvia Children's Hospital /Sahlgrenska University Hospital (SU), Sahlgrenska Academy, Dept of Pediatrics, University of Gothenburg
Locations (1):
- The Queen Silvia Children's Hospital / Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided